CLINICAL TRIAL: NCT00338780
Title: A Randomised, Double-Blinded, Placebo-Controlled Trial of Lamivudine Treatment in HBeAg Negative Chronic Hepatitis B Patients (in Asia)
Brief Title: Trial of Lamivudine Treatment in HBeAg Negative Chronic Hepatitis B Patients (in Asia)
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Chinese University of Hong Kong (Other)
Collaborators: GlaxoSmithKline (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: NUC30934
Record Dates: First submitted 2006-06-19; First posted 2006-06-20 (Estimated); Last update posted 2006-10-30 (Estimated); Status verified 2006-10

CONDITIONS: Chronic Hepatitis B
Keywords: Chronic Hepatitis B; Lamivudine; HBeAg negative
MeSH Terms: conditions — Hepatitis B, Chronic | interventions — Lamivudine

INTERVENTIONS:
Drug: Lamivudine/ Placebo 100mg daily

SUMMARY:
The aim is to investigate whether Lamivudine 100mg daily is effective in the long term treatment of HBeAg negative chronic HBV infected patients with active liver disease in Asia

DETAILED DESCRIPTION:
Recent studies have proved lamivudine a very potent antiviral drug in suppressing viral replication and improving hepatic necro-inflammation with minimal adverse effects in HBeAg positive chronic hepatitis B patients. The efficacy of lamivudine in HBeAg positivce Asian patients has been weel established. However, the evidence in HBeAg negative patients is limited.

In the absence of HBeAg seroconversion, guidance on the clinical management of HBeAg negative hepatitis B patitents treated with lamivudine and data on the efficacy of lamivudine in controlling pre-core HBV disease long-term is still needed. Existing data in HBeAg negative/ HBV DNA positive HBV demonstrate clear and statisticallysignificant serological benefit of lamivudine over placebo during treatment. Limited sustained response was observed post-treatment following a one year treatment period. Whether these results can be applied to patients in Asia is uncertain. This study is therefore intended to further assess te efficacy profile over an extended treatment period in the Asian population.

ELIGIBILITY:
Inclusion Criteria:

* Age=>18 years
* HBsAg positive and HBeAg negative for at least 6 months prior to screening
* Serum HBV-DNA postiviet, HBeAg negative and HBeAb positive at the same timepoint on at least one occasion during the last 6 months
* ALT >1.5 to 10 x upper limit of normal for at least two occasions within the previous 6 months and at screening, or ALT > upper limit normal and with at least one biochemical flare-up (ALT > 200IU/l) in the last 12 months.
* Informed writted consent
* Liver biopsy material/ slides taken within the previous 12 months, and at least 5 months after any previous antiviral treatment which show evidence of active liver disease (ie. evidence of necroinflammatory activity)
* Written informed consent

Exclusion Criteria:

* Hepatocellular carcinoma
* ALT > 10xULN at screening or history of acute exacerbation leading to transient decompensation
* Serum hepatitis C, hepatitis D or HIV
* Decompensated liver desease as indicated by any of the following: serum bilirubin >3mg/dL, prothrombin time >=2 seconds prolonged above upper limit of reference range, serum albumin <28g/L, history of variceal haemorrhage, presence of intractable ascites at the screening assessment.
* Encepalopathy
* Planned for liver transplantation or previous liver transplantation
* Evidence of autoimmune hepatitis
* Amylase and/ or lipase > 2 times upper limit of reference range
* Serum creatinine >1.5 times upper limit of reference range
* Haemoglobin < 11g/dL
* WBC count <3x10^9/L
* Platelets <100x10^9
* Serious concurrent medical illness other than hepatitis B
* Use of immunosuppressive therapy, immunomodylatory therapy or chronic antiviral thgerpay with other agents within the previous 6 months or during the study
* Previous treatment with lamivudine or famciclovir within the last 6 months
* History of hypersensitivity to nucleoside analogues
* Women of childbearing potential not practising adequate contraception
* Pregnancy or lactation
* Receipt of any investigational drug within 30 days of the first dose of study drug
* Child-Pugh class B or C cirrhosis

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Dates: Start 2000-11; Study Completion 2005-01

PRIMARY OUTCOMES:
Proportion of patients with complete response (normalisation of LAT, ie. <1xULN and disappearance of HBV DNA, lower limit of detection), at MOnth 24

SECONDARY OUTCOMES:
Proportion of patients with partial response
Histological improvement at month 24
Proportion of patients with complete response post-treatment (at Month 30)
Proportion of patinets with partial response post-treatment (at Month 30)
Progression of fibrosis
Progression of fibrosis to cirrhosis
HBsAg seroconversion
Safety of treatment

CONTACTS AND LOCATIONS:
Overall Officials: Joseph JY Sung, PhD, Principal Investigator — Chinese University of Hong Kong
Locations (1):
- Cheng Suen Man Shook Hepatitis Center, Institute of Digestive Disease, The Chinese University of Hong Kong, Prince of Wales Hospital, Hong Kong SAR, China

REFERENCES:
- [Background] Tassopoulos NC, Volpes R, Pastore G, Heathcote J, Buti M, Goldin RD, Hawley S, Barber J, Condreay L, Gray DF. Efficacy of lamivudine in patients with hepatitis B e antigen-negative/hepatitis B virus DNA-positive (precore mutant) chronic hepatitis B. Lamivudine Precore Mutant Study Group. Hepatology. 1999 Mar;29(3):889-96. doi: 10.1002/hep.510290321. PMID 10051494
- [Background] Maynard JE. Hepatitis B: global importance and need for control. Vaccine. 1990 Mar;8 Suppl:S18-20; discussion S21-3. doi: 10.1016/0264-410x(90)90209-5. PMID 2139281
- [Background] Tu H, Xiong SD, Trepo C, Wen YM. Frequency of hepatitis B virus e-minus mutants varies among patients from different areas of China. J Med Virol. 1997 Feb;51(2):85-9. doi: 10.1002/(sici)1096-9071(199702)51:23.0.co;2-n. PMID 9021537
- [Background] Tu H, Li PY, Wen YM. Anti-HBe titre in patients infected with wild-type and e-minus variant of hepatitis B virus. Res Virol. 1996 Jan-Feb;147(1):39-43. doi: 10.1016/0923-2516(96)80238-x. PMID 8882339
- [Background] ter Borg F, ten Kate FJ, Cuypers HT, Leentvaar-Kuijpers A, Oosting J, Wertheim-van Dillen PM, Honkoop P, Rasch MC, de Man RA, van Hattum J, Chamuleau RA, Reesink HW, Jones EA. Relation between laboratory test results and histological hepatitis activity in individuals positive for hepatitis B surface antigen and antibodies to hepatitis B e antigen. Lancet. 1998 Jun 27;351(9120):1914-8. doi: 10.1016/s0140-6736(97)09391-4. PMID 9654258
- [Background] Brunetto MR, Giarin MM, Oliveri F, Chiaberge E, Baldi M, Alfarano A, Serra A, Saracco G, Verme G, Will H, et al. Wild-type and e antigen-minus hepatitis B viruses and course of chronic hepatitis. Proc Natl Acad Sci U S A. 1991 May 15;88(10):4186-90. doi: 10.1073/pnas.88.10.4186. PMID 2034663
- [Background] Chu CM, Yeh CT, Chiu CT, Sheen IS, Liaw YF. Precore mutant of hepatitis B virus prevails in acute and chronic infections in an area in which hepatitis B is endemic. J Clin Microbiol. 1996 Jul;34(7):1815-8. doi: 10.1128/JCM.34.7.1815-1818.1996. PMID 8784599
- [Background] Chan HLY, Hui Y, Ching JYL, Leung NWY, Chan FKL, Sung JJY. Can we predict disease activity in chronic hepatitis B virus (CHB) infected patients with negative HBeAg. Gastroenterology 1999; 116: A1195
- [Background] Chan HLY,Ghany MC, Lok ASF. Hepatitis B. In Schiff ER, Sorrell MF, Madrey WC, Eds. Schiff's Deseases of the LIver, 8th ed. Lippincott-Raven Publishers, New York, 1998:757-92
- [Background] Zaaijer HL, ter Borg F, Cuypers HT, Hermus MC, Lelie PN. Comparison of methods for detection of hepatitis B virus DNA. J Clin Microbiol. 1994 Sep;32(9):2088-91. doi: 10.1128/jcm.32.9.2088-2091.1994. PMID 7814529
- [Background] Laras A, Koskinas J, Avgidis K, Hadziyannis SJ. Incidence and clinical significance of hepatitis B virus precore gene translation initiation mutations in e antigen-negative patients. J Viral Hepat. 1998 Jul;5(4):241-8. doi: 10.1046/j.1365-2893.1998.00109.x. PMID 9751010
- [Background] Chan HL, Hussain M, Lok AS. Different hepatitis B virus genotypes are associated with different mutations in the core promoter and precore regions during hepatitis B e antigen seroconversion. Hepatology. 1999 Mar;29(3):976-84. doi: 10.1002/hep.510290352. PMID 10051506
- [Background] Krajden M, Minor J, Cork L, Comanor L. Multi-measurement method comparison of three commercial hepatitis B virus DNA quantification assays. J Viral Hepat. 1998 Nov;5(6):415-22. doi: 10.1046/j.1365-2893.1998.00129.x. PMID 9857351
- [Background] Lai VC, Guan R, Wood ML, Lo SK, Yuen MF, Lai CL. Nucleic acid-based cross-linking assay for detection and quantification of hepatitis B virus DNA. J Clin Microbiol. 1999 Jan;37(1):161-4. doi: 10.1128/JCM.37.1.161-164.1999. PMID 9854083
- [Background] Chan HLY, Leung NY, Lau TCM, Wong ML, Sung JJY. Comparison of three different hepatitis B virus (HBV) DNA assays in monitoring of anti-viral therapy. Hepatology 1999 (in press)